CLINICAL TRIAL: NCT02598479
Title: The IPTLD QoL Broad Study A Quality of Life Study Using Insulin Potentiation Targeted LowDose (IPTLD) Chemotherapy and Nutrition Therapy in the Treatment of Cancer
Brief Title: A Quality of Life Study Using Insulin Potentiation Targeted LowDose (IPTLD) Chemotherapy and Nutrition Therapy in the Treatment of Cancer
Acronym: IPTLDAZCAM
Status: Withdrawn | Type: Observational
Why Stopped: The IRB which was overseeing the study stopped overseeing it
Sponsor: Best Answer for Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol V1- 08-12-2015
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Cancer
Keywords: Cancer; Insulin Potentiation Low Dose Chemotherapy; IPT; IPTLD; Nutrition therapy
MeSH Terms: conditions — Neoplasms | interventions — Nutrition Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IPTLD and nutrition therapy: Patients presenting to the Arizona Center for Advanced Medicine for the treatment of cancer using Insulin Potentiation Low Dose Chemotherapy and Nutrition Therapy
  Interventions: Other: IPTLD and nutrition therapy

INTERVENTIONS:
Other: IPTLD and nutrition therapy — The measurement of Quality of Life in patients who choose to use Insulin Potentiation Low Dose Therapy and Nutritional Therapy in the treatment of cancer

SUMMARY:
The IPTLD QoL Broad Study.

DETAILED DESCRIPTION:
A Quality of Life Study Using Insulin Potentiation Targeted LowDose (IPTLD) Chemotherapy and Nutrition Therapy in the Treatment of Cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cancer,
* age older than 18 years,
* requesting IPTLD and nutrition therapy

Exclusion Criteria:

* diagnosis other than cancer,
* age younger than 18 years,
* requesting conventional chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who have chosen to receive IPTLD with nutrition therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Quality of Life measured by questionnaires | 5 years
  Improvement in Quality of Life using Insulin Potentiation Low Dose Chemotherapy and Nutrition Therapy for the Treatment of Cancer, as measured by MD Anderson's MDASI questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Martha M Grout, MD, MD(H), Principal Investigator — Arizona Center for Advanced Medicine
Locations (1):
- Arizona Center for Advanced Medicine, Scottsdale, Arizona, United States